CLINICAL TRIAL: NCT05020808
Title: The Effect of a Plant Protein Isolate on Muscle Protein Synthesis in Humans at Rest, and After Resistance Exercise: A Randomized Controlled Trial
Brief Title: The Effect of a Plant Protein Isolate on Muscle Protein Synthesis in Humans at Rest and After Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Marigot Ltd. (Industry); Enterprise Ireland (Other Government)
Responsible Party: Principal Investigator, Robert Davies, Principal Investigator, University of Limerick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020_04_07_EHS
Record Dates: First submitted 2021-08-17; First posted 2021-08-25 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Metabolism; Exercise; Dietary Supplements
Keywords: amino acids; deuterium oxide; humans; protein synthesis; plant proteins; resistance training; skeletal muscle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Block randomized control trial, parallel group design
Who Masked: Participant
Masking Description: Single blind (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nonessential amino acid formulation (NEAA) (Sham Comparator): Novel non-essential amino acid blend dosed at 0.33 g/kg body mass in 400 ml of water. Postprandial muscle protein synthesis at rest, and after resistance exercise to be measured by deuterium incorporation in to skeletal muscle sampled by bilateral microbiopsies.
  Product Number: NEAA56812
  Interventions: Dietary Supplement: NEAA
- Plant Protein Isolate (PPI) (Active Comparator): Plant protein isolate (Fava bean) dosed at 0.33 g/kg body mass in 400 ml of water. Postprandial muscle protein synthesis at rest, and after resistance exercise to be measured by deuterium incorporation in to skeletal muscle sampled by bilateral microbiopsies.
  Product Number: FP2011273
  Interventions: Dietary Supplement: PPI

INTERVENTIONS:
Dietary Supplement: NEAA — Food grade mixture of non-essential amino acids in powdered form to be dissolved in water. Supplied by Marigot Ltd, Cork, Ireland
  Arms: Nonessential amino acid formulation (NEAA)
Dietary Supplement: PPI — Food grade plant (legume - Fava) protein isolate to be dissolved in water. Supplied by Marigot Ltd, Cork, Ireland
  Other Names: Plant Protein Isolate
  Arms: Plant Protein Isolate (PPI)

SUMMARY:
Plant-based proteins contain several amino acids that are essential to signal growth, reconditioning, maintenance and preservation of skeletal muscle mass. This study aims to inform on the nutrient activation of muscle protein synthesis (MPS) by feeding a plant protein isolate equivalent to 0.33 g of protein per kilogram of body mass.

DETAILED DESCRIPTION:
Participants: 32 young, healthy men and women aged 18 - 35 years. Intervention: Plant protein isolate (PPI) and nonessential amino acid control (NEAA) Study Design: Block randomised control trial. Two group parallel design. Primary outcome: Myofibrillar fractional synthetic rate (myoFSR).

Preliminary screening/familiarization consists of: medical history, dietary assessment and examination by a medical doctor and a qualified dietician, blood sample to be evaluated for health-related contraindications, body composition measurement by dual energy x-ray absorptiometry (DXA), isokinetic knee extensor strength tests.

Pre-trial: A metered dose of deuterium oxide (5ml/kg) will be ingested and blood and/or saliva (~5ml) samples will be collected pre/post ingestion.

Experimental trial: Blood, saliva and bilateral m.vastus lateralis microbiopsies (~100 mg) collected. A unilateral resistance-training session consisting of knee extensor contractions will be completed. Following exercise cessation participants will ingest 0.33 g/kg body mass of either: a nonessential amino acid formulation or a plant-protein isolate. A saliva sample and a 2nd set of bilateral m.vastus lateralis microbiopsies are collected 3 h postingestion.

ELIGIBILITY:
Inclusion Criteria:

- Men and women aged 18 to 35 years

Exclusion Criteria:

* Known intolerance to any item contained in the protein products.
* Blood borne disease risk, current illness or medication that would adversely affect participation
* Known adverse reaction to venepuncture and/or biopsy
* Inability to undertake resistance exercise
* Inability to adhere to protocol guidelines

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Myofibrillar fractional synthetic rate change | 4 hours
  The fractional rate of myofibrillar protein synthesis measured by deuterium incorporation into skeletal muscle sampled by microbiopsy

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Jakeman, PhD, Principal Investigator — University of Limerick; Robert W Davies, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No